CLINICAL TRIAL: NCT01756976
Title: Clinical Evaluation of the OrthoPAT Advance System
Status: Completed | Type: Observational
Sponsor: Haemonetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: TP-CLN-100257
Record Dates: First submitted 2012-11-26; First posted 2012-12-28 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Transmission, Blood, Recipient/Donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Investigational Device: The 510k cleared OrthoPAT Advance will be used in this standard of care arm.
  Interventions: Device: OrthoPat Advance
- Control Group: The commercially available OrthoPAT will be used in this arm. This is an observational trial and there is no intervention.

INTERVENTIONS:
Device: OrthoPat Advance — The device will be used initially in hysterectomy procedures. After a confirmation of product quality, the device will be used in routine orthopedic procedures.
  Groups: Investigational Device

SUMMARY:
This study is intended to provide additional performance data of the OrthoPAT Advance in routine orthopedic surgery.

DETAILED DESCRIPTION:
The OrthoPAT Advance system is being developed by Haemonetics to change the user interface, especially for adding calculations for Estimating Blood Loss- (EBL). The OrthoPAT® serves as the predicate device. The following items will be changed in the OrthoPAT Advance system compared to OrthoPAT:

* Software & User Interface - ability to enter irrigant and anti-coagulant volumes and allow Estimated Blood Loss (EBL) calculation to be made by OrthoPAT Advance.
* Hardware -

  * Redesign of reservoir and filter to process blood earlier by reducing hold-up volume and improve fluid visualization in reservoir.
  * Extended battery life.

It is not intended to validate the major changes in the OrthoPAT Advance device (reservoir / filter and EBL), which will be conducted as lab based tests. The correct functioning of the reservoir / filter and EBL changes will be confirmed in the clinical setting in this study. However the most rigorous challenge to the filter will be by presenting the worst case media and this can only be controlled in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 18 years
* Subject is scheduled for a total knee/hip replacement/ revision or a hysterectomy.
* Subjects determined eligible per site standard of care for use of intra- and post-operative use of cell salvage device

Exclusion Criteria:

For subjects where product is transfused

* Subject is undergoing a trauma procedure where there is a possibility of contamination from an open wound.
* Patient is diagnosed with sepsis.
* Patient is diagnosed with sickle-cell anemia.
* Malignant cells may be mixed with blood salvaged from the surgical field.
* Prostatic or amniotic fluid is mixed with blood salvaged from the surgical field.
* Blood salvaged from the surgical field may be contaminated from an active infection at wound/drain site.
* Blood salvaged from the surgical field contains topical hemostatic agents, anti-bacterial agents, or wound irrigants not intended for parenteral use.

For all subjects:

* Subject is undergoing a procedure which involves high, rapid blood loss such as liver transplants, certain cardiovascular procedures, and trauma procedures where blood loss is high (per Investigators judgment).
* Any procedure terminated prior to completion by subject request, operator decision or error, or device error.
* Any subject with which at least 200mL of filtered blood or 1 full disc is not available for processing and data collection within the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects scheduled for hysterectomy or orthopediac procedures.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2012-12; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Waters, MD, Principal Investigator — University of Pittsburgh Medial Center
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device | Control Group
Started | 76 | 8
Completed | 73 | 8
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Investigational Device | Control Group | Total
Number analyzed (Participants) | 76 | 8 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 8 | 66
  >=65 years | 18 | 0 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (19) | 46 (9) | 55 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 8 | 60
  Male | 24 | 0 | 24
Region of Enrollment [Number; unit: participants]
  United States | 76 | 8 | 84

OUTCOME MEASURES:

1. Primary Outcome: Washed RBC Hematocrit
Description: The Hematocrit of the RBC shall be > 50%.
Time Frame: < 4 hours
Measure: Mean (Standard Deviation); unit: percentage of HcT
Arm/Group | Investigational Device | Control Group
Number analyzed (Participants) | 15 | 6
percentage of HcT | 55.43 (7.47) | 56.48 (5.28)

ADVERSE EVENTS:
Arm/Group | Investigational Device | Control Group
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/8
Other Adverse Events (participants affected / at risk) | 0/73 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less